CLINICAL TRIAL: NCT04198558
Title: A Randomised, Double-blind, Placebo-controlled Study of the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of MEDI0618 in Healthy Male and Female Volunteers
Brief Title: A Study of the Safety, Tolerability and Pharmacokinetics of MEDI0618 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D7060C00001; 2019-002128-33 (EudraCT Number)
Record Dates: First submitted 2019-11-25; First posted 2019-12-13 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Chronic Pain
Keywords: Double-blind; Placebo-controlled; Safety and Tolerability Study; Healthy Volunteers
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Dose Level 1 (Experimental): MEDI0618 or placebo
  Interventions: Drug: MEDI0618; Drug: Placebo
- Dose Level 2 (Experimental): MEDI0618 or placebo
  Interventions: Drug: MEDI0618; Drug: Placebo
- Dose Level 3 (Experimental): MEDI0618 or placebo
  Interventions: Drug: MEDI0618; Drug: Placebo
- Dose Level 4 (Experimental): MEDI0618 or placebo
  Interventions: Drug: MEDI0618; Drug: Placebo
- Dose Level 5 (Experimental): MEDI0618 or placebo
  Interventions: Drug: MEDI0618; Drug: Placebo
- Dose Level 6 (Experimental): MEDI0618 or placebo
  Interventions: Drug: MEDI0618; Drug: Placebo
- Dose Level 7 (Experimental): MEDI0618 or placebo
  Interventions: Drug: MEDI0618; Drug: Placebo
- Dose Level 8 (Experimental): MEDI0618 or placebo
  Interventions: Drug: MEDI0618; Drug: Placebo
- Dose Level 9 (Experimental): MEDI0618 or placebo
  Interventions: Drug: MEDI0618; Drug: Placebo

INTERVENTIONS:
Drug: MEDI0618 — MEDI0618 A novel human immunoglobulin antibody
Drug: Placebo — Placebo

SUMMARY:
This is a randomised, placebo-controlled study of the safety and tolerability of single doses of MEDI0618 in healthy volunteer subjects.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled study of the safety, tolerability and pharmacokinetics of single ascending doses of MEDI0618 in healthy male and female volunteers.

This study will include 9 planned cohorts; 8 cohorts will receive single ascending doses of MEDI0618 or placebo by intravenous administration, 1 cohort will receive MEDI0618 or placebo by subcutaneous administration.All subjects will undergo scheduled safety, tolerability, pharmacokinetic and immunogenicity assessments while in the clinical unit and as outpatients to the end of the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women of non-childbearing potential aged 18 to 55 years
* Normal 12-lead ECG at screening and on day of dosing
* Physical examinations with no significant findings at screening
* Be able to understand and comply with protocol requirements

Exclusion Criteria:

* Participation in another clinical study with an investigational product (IP) within half-lives of the IP or 3 months, whichever is longer, prior to screening
* Requires treatment with another biological therapeutic agent
* Inability to comply with study-related requirements
* History of severe allergy or hypersensitivity reactions
* History of significant psychiatric disorder
* Presence of any clinically significant illness
* History of cancer
* Any clinically important abnormality physical examination, vital signs, ECG or laboratory test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 85 days
  Adverse Events
Incidence of Treatment-Emergent Serious Adverse Events | Up to 85 days
  Serious Adverse Events
Vital Signs | Up to 85 days
  Heart Rate in beats per minute
Vital Signs | Up to 85 days
  Blood pressure in mm Hg
Body Weight | Up to 85 days
  Weight in kg
Height | Up to 85 days
  Height in meters Height and weight will be combined to report BMI in kg/m^2
Clinical Chemistry | Up to 85 days
  Measurement of Albumin, Protein, Aspartate transaminase, Alanine transaminase, Alkaline phosphatase, Bilirubin, Calcium, Creatine phosphokinase, C-reactive protein, Glucose, Blood urea nitrogen, Phosphate, Potassium, Sodium, Chloride and Bicarbonate
Haematology | Up to 85 days
  Measurement of Haemoglobin, Haematocrit, Leukocyte count, Platelet count, Erythrocyte count, Reticulocyte count, Mean corpuscular haemoglobin
Thyroid Function | Up to 85 days
  Measurement of Thyroid-stimulating hormone and free thyroxine
Renal Function | Up to 85 days
  Measurement of Glomerular filtration rate
Urinalysis | Up to 85 days
  Measurement of Haemoglobin, Leukocytes, Glucose, Protein and Creatinine
12-Lead Electrocardiogram | Up to 85 days
  Measurement of Heart rate; PR, QRS, RR, QT and QTc intervals from digital recordings
Physical Examination | Up to 85 days
  General physical examination

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | Up to 85 days
  Peak concentration of MEDI0618 in plasma
Time to maximum concentration (tmax) | Up to 85 days
  Time to maximum concentration of MEDI0618 in plasma
Area under the concentration versus time curve (AUC) | Up to 85 days
  Calculated area under the concentration versus time curve for MEDI0618
Terminal half-life | Up to 85 days
  Time required for the plasma concentration of MEDI0618 to decrease by 50%
Bioavailability | Up to 85 days
  The fraction of MEDI0618 administered that is available to the systemic circulation

OTHER OUTCOMES:
Anti-drug antibody incidence and titres | Up to 85 days
  Anti-drug (MEDI0618) antibody incidence and titres

CONTACTS AND LOCATIONS:
Overall Officials: Tharani Chessell, PhD, Study Director — AstraZeneca; Stanislav Ignatenko, Medical Doctor, Principal Investigator — Charite Research Organisation
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual patient-level data will be shared.
Time Frame: After CSR sign-off.
Access Criteria: Qualified researchers.

REFERENCES:
- See also: CSR SYNOPSIS — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7060C00001&attachmentIdentifier=a34c53be-52e3-4161-9a92-fec1c1c2e7f1&fileName=CSR_SYNOPSIS_D7060C00001_Version_1.0_final-synopsis-Redacted_06Mar2023.pdf&versionIdentifier=